CLINICAL TRIAL: NCT02703506
Title: Effectiveness of a Pain Education Program on Chronic Neck Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OE22/2015
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental. Pain Education Program (Experimental): Ten group sessions of treatment with a patient education pain for chronic neck pain (biopsychosocial approach). The group sessions of 60-120 minutes twice a week with a maximum of 10 participants.
  Interventions: Other: Session of Pain Education programe
- Control (Active Comparator): The control group: individualized session of physical therapy (TENS and exercise).
  Five individual sessions twice a week, will be performed of transcutaneous electrical nerve stimulation (TENS) on neck area an exercises .
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Session of Pain Education programe — Five group sessions of patient education pain of 60-120 minutes one for week with a maximum of 10 participants.
  Arms: Experimental. Pain Education Program
Other: Control Group — Five individual sessions twice a week, will be performed of transcutaneous electrical nerve stimulation (TENS) on neck area an exercises
  Arms: Control

SUMMARY:
This project aims to study the effectiveness of a pain education program in the improvement of chronic pain and disability/impairment. Assuming the definition established in the United States in 1975 on the fourth working group of the National Conference on Preventive Medicine: "Health education must be a process that informs, motivates and helps people to adopt and maintain practices and healthy lifestyles, environmental advocates changes necessary to facilitate these objectives and professional training and directs research towards the same objectives. " Once the need of educating patients is stablished on subjects with diseases, it is necessary to encourage them to actively participate on the control of them and to achieve significant improvement of adherence

DETAILED DESCRIPTION:
BACKGROUND AND PURPOSE:

Patient education over the knowledge of pain causes and perpetuating psicosocial factos, so as a gradual physical therapy intervention may success in modifying habits, and consequently emotional state and behaviour in order to maintain or recover subject's social participation being this program effective in pain diminution over chronic neck pain.

Main goal: To evaluate the effectiveness of a pain education program for patients with chronic neck pain, to decrease the intensity of pain in front of one physiotherapy program (TENS and exercise)

Experimental group: Will receive five group sessions of 60-120 minutes twice a week with a maximum of 10 participants.

Control group: Five individual sessions twice a week, will be performed of transcutaneous electrical nerve stimulation (TENS) on neck area an exercises.

OUTCOMES

Primary outcome

* Intensity of pain, measured by the visual analog scale: VAS. The mean of the values wil be calculated described in the assessment, the mean of the last week was also compiled.
* The degree of neck disability/impairment measured using the Northwick Park Pain Questionnaire (NPPQ)

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old
* Subjects diagnosed with chronic neck pain.

Exclusion Criteria:

* Patients with acute and subacute neck pain. Those presenting inflammatory, neurologic, rheumatic or heart disease or pacemakers. Patients with severe osteoporosis, fractures, dislocations, vertebrobasilar insufficiency, infection, metastatic tumor, pre and post-surgical etiology recent (less than one year after the intervention).

Psychopathology patients diagnosed by their doctor. Subjects who do not understand or speak the Spanish language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change From Baseline in Pain Scores on the Visual Analog Scale at three months
  Measured by a Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel PM Pecos-Martín, Dr, Study Director — Alcala University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Munoz M, Rodriguez-Costa I, Lebrijo-Perez G, Pecos-Martin D, Gallego-Izquierdo T, Perez-Martin Y. Design of a Health Education Program to Manage Chronic Neck Pain: Protocol for a Development Study. JMIR Res Protoc. 2024 Oct 1;13:e56632. doi: 10.2196/56632. PMID 39353191